CLINICAL TRIAL: NCT02199834
Title: A Quality Improvement Project Evaluating the Effect of Regular Personalized Feedback Report and Peer Support for Patients With Diabetes in Hong Kong
Brief Title: Effect of Personalized Feedback Report and Peer Support on Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Junmei YIN, Ms., Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CRE-2013.033
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes
Keywords: diabetes; peer support; personalized feedback report
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Peer group (Experimental): 24 patients who have good glycemic control and self-care will be trained as peer supporters to deliver peer support to this group under supervision by a program manager. Peer supporters will call their peers at least 12 times a year to provide both informational and emotional support. Half of the patients in this group will be randomized to receive a personalized feedback report displaying trends of metabolic control of A1c, BP, LDL-C, and body weight, with automated decision support based on their own attained values every 4 months through mails.
  Interventions: Behavioral: Peer support; Behavioral: Personalized feedback report
- Refused peer group (Other): Patients who fit the criteria of peers but refuse to be contacted by peer supporters will be signed as refused group. Half of the patients in this group will be randomized to receive a personalized feedback report displaying trends of metabolic control of A1c, BP, LDL-C, and body weight, with automated decision support based on their own attained values every 4 months through mails.
  Interventions: Behavioral: Personalized feedback report
- Report group (Experimental): Patients in this group will receive a personalized feedback report displaying trends of metabolic control of A1c, BP, LDL-C, and body weight, with automated decision support based on their own attained values twice a year through mails.
  Interventions: Behavioral: Personalized feedback report
- Usual care (No Intervention): Patients will receive standard usual care with clinicians' follow-up and referral with education to diabetes nurses if deemed necessary at in-charge clinicians' discretion.

INTERVENTIONS:
Behavioral: Peer support — 15 patients who have good glycemic control and self-care will be trained as peer supporters to deliver peer support under supervision by a program manager. Peer supporters will call their peers at least 12 times a year to provide both informational and emotional support.
  Arms: Peer group
Behavioral: Personalized feedback report — Patients will receive a personalized feedback report displaying trends of metabolic control of A1c, BP, LDL-C, and body weight, with automated decision support based on their own attained values every 4 months through mails.
  Arms: Peer group; Refused peer group; Report group

SUMMARY:
In this project, the investigators hypothesize that in an integrated, multifaceted, team-based program incorporating comprehensive assessment with risk stratification, diabetic patients with high risk of negative emotions and hospitalization will benefit from additional peer support which will improve their psychological health, cardio-metabolic control, self-management, quality of life and reduce hospitalization. The investigators further hypothesize that peer support will interact with regular personalized feedback reporting to improve clinical outcomes.

DETAILED DESCRIPTION:
Diabetes self-management is often emotionally and physically taxing, demanding lifelong commitment to medication adherence and lifestyle modification. People with diabetes have to be well-educated and supported to make clinical decisions in their daily living. However, most diabetes self-management education (DSME) interventions are short-term and have little external support. In order to empower patients to self-manage over a lifetime after the initial DSME, ongoing multidisciplinary programs which coordinates individual components of care into a structured system and further supported by reinforcement through multiple contacts are necessary to provide practical tips as well as social and psychological support to diabetic patients, so as to sustain behavioral changes and improve metabolic control.

Based on these principles, the Joint Asia Diabetes Evaluation (JADE) Program was developed in 2007 as a quality improvement initiative to deliver technologically integrated and multidisciplinary team-based care. It is enabled by a web-based portal containing templates which guide care providers in providing standardized comprehensive assessments, the results of which are then used for personalized risk stratification and feedback reports. The personalized feedback report contains the patient's risk category according to the JADE definition, with visual displays of important trends including those of glycated haemoglobin (HbA1c), blood pressure (BP), low-density-lipoprotein-cholesterol (LDL-C), and body mass index (BMI), and practical suggestions to help the individual to reach multiple treatment targets based on the latest values.

On the other hand, according to a recent WHO consultation report, peer support intervention is considered to have enormous potential to improve self-management in patients with chronic disease. Programs using peer supporters to teach and support their peers with diabetes have shown significant reductions in HbA1c, enhanced self-efficacy, improved health status and better self-management behaviors. In our previous study, we found that a combined program which integrates structured care, peer support and clinical decision support by regular follow up report significantly improved psychological health and medication adherence of diabetic patients, and reduced hospitalization of patients with negative emotions like depression, distress, and anxiety, who were most likely to suffer from chronic kidney disease or poor glycemic control. In this program, we hypothesize that using a multifaceted program which incorporates structured care, personalized feedback reporting, and peer support to influence and motivate diabetic patients with high risk of hospitalization and negative emotions on diabetes self-management, will further improve their self-management, psychological health and metabolic control, and reduce hospitalization. We further hypothesize that receiving personalized feedback report with decision support will improve glycemic control and reduce hospitalization in patients with diabetes.

Around 286 patients with high risk of negative emotion and hospitalization will be invited to join the peer support program. We anticipate that half of the patients will agree (n=143) and be assigned 24 peer supporters on a 5~6:1 ratio. Peer supporters are patients who have good glycemic control and self-care and trained to provide both informational and emotional support to the peer group. For patients who decline to participate, they will be identified as refused peer group and their reasons for declining will be documented. Half of the patients in each group will be randomized to receive 2 personalized feedback reports through the mail.

1200 adult patients consecutively enrolled in JADE program will be recruited and half of them (n=600) will be randomized to receive a personalized feedback report twice a year. All patients will be followed up at their usual clinics and will be observed for at least 1 year when we shall evaluate the effects of providing regular personalized report on clinical outcomes including metabolic control and hospitalization.

To evaluate the independent effects of peer support , we further used a case-control design to. Within the 1200 patients who were not offered peer support, a group of patients who met the criteria of "high risk" were matched to those agreed to receive peer support on a 3:1 basis by age, gender, diabetes duration, and baseline HbA1c as a control group. Data of metabolic control and hospitalization of the control group were retrieved from the CMS and compared to that of the peer group after 1 year.

The study objectives are:

1. To study the effect of regular personalized feedback reports to patients with diabetes managed within an integrated care program on hospitalization and metabolic control, irrespective of their risk levels.
2. To study the feasibility of using trained diabetes patients (peer supporters) to assist diabetes educators in diabetes management.
3. To study the acceptability of peer support in a real life setting and the effects of non-participation in peer support program on clinical outcomes including hospitalization and glycemic control in high risk patients for negative emotions and multiple risk factors.
4. To study the independent and interactive effects of peer support and regular personalized feedback report on cardio-metabolic risk factor control, psychological health, self-efficacy, self-management, quality of life and hospitalization rates in patients with diabetes at high risk for negative emotions and multiple risk factors.

ELIGIBILITY:
Inclusion Criteria:

For peer supporters:

* Patients with type 2 diabetes.
* Aged between 18 and 75 years (inclusive).
* Chinese ethnicity.
* Stable glycemic control (HbA1c<7.5%) and self-rated health status≥80 as assessed by EQ5D visual scale.
* Enthusiastic and willing to become peer supporters.

For peers:

* Patients with diabetes.
* Aged between 18 and 75 years (inclusive).
* Chinese ethnicity.
* At least 1 of the following risk factors: HbA1c≧8%/ BMI≧27.5 kg/m2/ Waist circumstance≧80cm in women or ≧90cm in men/ Chronic kidney disease (CKD) defined as estimated glomerular filtration rate less than 60 ml/min /1.73m2.
* Agree to receive peer support

For report group and usual care group:

* All Chinese diabetes patients between 18-75 years of age who undergo comprehensive assessment and join the JADE program.

Exclusion Criteria:

For peer supporters:

* HbA1c≧7.5% in last 6 months.
* Terminal malignancy or other life-threatening diseases.
* Unstable mental diseases.
* Unable to communicate in Chinese.

For peers:

* Terminal malignancy or other life-threatening diseases.
* Unstable mental illness.
* Unable to communicate in Chinese.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1488 (Actual)
Dates: Start 2013-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Hospitalization | 12 months
  The number of, and the corresponding reasons for hospital admissions, using the International Classification of Diseases-9th version in the discharge summary, retrieved from the Hong Kong Hospital Authority Central Computer System.
Change of HbA1c | 12 months

SECONDARY OUTCOMES:
Changes in self-efficacy | 12 months
  Diabetes Empowerment Scale (DES)
Change in cardio-metabolic risk factors | 12 months
  Absolute change in risk factors (A1c, LDL-C, body weight, blood pressure)
Clinically meaningful reductions in risk factors | 12 months
  Percentage of patients with clinically meaningful reductions in risk factors (A1c >=0.5%; LDL-C>=30%; systolic BP>=10 mmHg and body weight>=3% compared with baseline)
Percentage of patients attaining multiple treatment goals | 12 months
  Percentage of patients attaining multiple treatment goals (A1c <7%, LDL-C<2.6 mmol/L and BP<130/80 mmHg).
Satisfaction survey by participants | 12 months
  Satisfaction survey by peers
Change in negative emotions | 12 months
  Depression Anxiety Stress Scale-21 (DASS21)
Change in quality of life | 12 months
  WHO Quality of Life-Bref (WHOQOL-BREF),
Change in health-related quality of life | 12 months
  Euro Quality of Life (EQ5D)
Change in depressive symptom | 12 months
  Patient Health Questionnaire (PHQ9).

CONTACTS AND LOCATIONS:
Overall Officials: Junmei YIN, MPH, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong SAR, China